CLINICAL TRIAL: NCT04428099
Title: Effectiveness of a Healthy Lifestyle Promotion Program as Adjunctive Teletherapy for Treatment-resistant Major Depression During Covid 19 Pandemic: A Randomized Clinical Trial Protocol
Brief Title: Healthy Lifestyle Promotion as Adjunctive Teletherapy for Treatment-resistant Major Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMD01
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: heallthy Lifestyle; Minfullness based cognitive therapy; Teletherapy
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Lifestyle change promotion program
  Interventions: Behavioral: Lifestyle change promotion program; Behavioral: Written Information
- Control 1 (Active Comparator): MBCT program
  Interventions: Behavioral: Mindfullness based cognitive program; Behavioral: Written Information
- Control 2 (Placebo Comparator): Usual care
  Interventions: Behavioral: Written Information

INTERVENTIONS:
Behavioral: Lifestyle change promotion program — The intervention consists of 8 group sessions centered on healthy physical activity, healthy diet, social life, Good Sleep Hygiene, healthy sun exposure, nature contact, how to stop ruminating, review and maintenance tips.
  Arms: Intervention
Behavioral: Mindfullness based cognitive program — The intervention consists of 8 group sessions with a mindfulness-based cognitive program
  Arms: Control 1
Behavioral: Written Information — Written information about lifestyle change suggestions

SUMMARY:
The main objective of the study will be to evaluate the effectiveness of an adjuvant lifestyle-based intervention for treatment-resistant patients with major depressive disorder. Patients will be allocated to one of these three groups: 1)Treatment prescribed by their mental health team plus written lifestyle change suggestions 2)Treatment prescribed by their mental health team plus written lifestyle change suggestions plus 8-week Mindfulness-based cognitive therapy (MBCT) program 3) Treatment prescribed by their mental health team plus written lifestyle change suggestions plus 8-week lifestyle change promotion program. We will collect patient data using the questionnaires administered at baseline, immediately after the intervention, and at six and 12-month follow-up. The primary outcome will be depression severity and secondary outcomes will include health-related quality of life.

DETAILED DESCRIPTION:
Depression is a very prevalent, incapacitating illness. The treatment available (psychotherapy and drug therapy) do not always manage to achieve complete remission of the symptoms or prevent its relapses or recurrences. For that reason, it is still necessary to investigate new adjuvant therapeutic antidepressant alternatives, especially if they can add efficacy to the treatment without reducing tolerance and safety. In the last few years, data have been growing about the usefulness of having patients who are depressed make specific changes in their lifestyles.

The main objective of the study will be to evaluate the effectiveness and efficiency of an adjuvant lifestyle-based intervention for treatment-resistant patients with major depressive disorder. Patients will be allocated to one of these three groups: 1)Treatment prescribed by their mental health team plus written lifestyle change suggestions 2)Treatment prescribed by their mental health team plus written lifestyle change suggestions plus 8-week MBCT program 3) Treatment prescribed by their mental health team plus written lifestyle change suggestions plus 8-week lifestyle change promotion program. Two control groups were designed: placebo-control (written lifestyle change suggestion) and active-control (MBCT). We selected this adjuvant therapy because MBCT has shown positive results as an adjunctive treatment for resistant depression in previous studies and it could be administered in a similar format as our intervention (8-weeks lifestyle change promotion program). We hypothesize that the lifestyle change promotion program at 12 months of follow-up will be more effective because patients will have better adherence to this intervention than to MBCT.

This study will be carried out during the COVID-19 pandemic, therefore the administration of the intervention will be administered by teletherapy. Different ways and technologies will be used to contact participants remotely: telephone calls, text messages, WhatsApp groups, and teleconferences.

We will collect patient data using the questionnaires administered at baseline, immediately after the intervention, and at six and 12-month follow-up. The primary outcome will be measured using the Beck Depression Inventory-II (BDI-II). Secondary outcomes will include Clinical Global Impressions (CGI) Scale, to quantify and track patient progress and treatment response over time and Health-related quality of life measured using the European Quality of Life-5 Dimensions Questionnaire (EQ-5D).

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or older.
* Diagnosis of Major Depressive Disorder as stated by the DSM-5.
* Two previous treatment failures (non-response to an adequate dose of potentially effective medication for an adequate length of time or treatment intolerance or refusal) in the current episode.
* At least one month of treatment with a psychiatrist and/or psychologist in the current episode.
* Physical and cognitive aptitudes to understand and give written informed consent.

Exclusion Criteria:

* Comorbidity with other medical conditions which would affect the Central Nervous System (CNS).
* Other severe psychiatric disorders (except for anxiety disorders or personality disorders)
* Other non-controlled severe medical diseases, infectious or degenerative which would interfere with affective symptomatology or the adherence to the hygienic-dietary recommendations.
* Patients with delusions or hallucinations which are congruent or non-congruent with mood.
* Patients with an important risk for suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-01-12 (Estimated); Study Completion 2022-07-12 (Estimated)

PRIMARY OUTCOMES:
Depression severity | 12 month
  Beck Depression Inventory-II (BDI-II)

SECONDARY OUTCOMES:
Health-related quality of life | 12 month
  Questionnaire (EQ-5D)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Illes Balears, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Derived] Navarro C, Yanez AM, Garcia A, Segui A, Gazquez F, Marino JA, Ibarra O, Serrano-Ripoll MJ, Gomez-Juanes R, Bennasar-Veny M, Salva J, Olivan B, Roca M, Gili M, Garcia-Toro M. Effectiveness of a healthy lifestyle promotion program as adjunctive teletherapy for treatment-resistant major depression during COVID 19 pandemic: A randomized clinical trial protocol. Medicine (Baltimore). 2020 Nov 6;99(45):e22958. doi: 10.1097/MD.0000000000022958. PMID 33157937